CLINICAL TRIAL: NCT02051634
Title: Efficacy of Fermented Papaya Preparation on Markers of Systemic Inflammation
Brief Title: Papaya Study ID:20140628
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Osato Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB20140628
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Systemic Inflammation; Aging
Keywords: Aging; Papaya; Fermented Papaya; Inflammation; Phytochemicals; Physical function; Quality of life; Fatigue; Health
MeSH Terms: conditions — Inflammation; Fatigue | interventions — fermented papaya preparation; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fermented Papaya Preparation (FPP) (Active Comparator): A total of 9 grams of FPP per day (divided into three 3 gram doses) will be consumed for 8 weeks. Participants will consume three 3g sachets containing FPP per day - once 30-40 min before breakfast, once 30-40 min before lunch, and once 30-40 min before dinner. Participants will open the sachet, empty contents into their mouth, and let it dissolve before swallowing.
  Interventions: Drug: Fermented Papaya Preparation (FPP); Drug: Sugar Pill
- Sugar Pill (Placebo Comparator): A total of 9 grams of placebo (sugar) per day (divided into three 3 gram doses) will be consumed for 8 weeks. Participants will consume three 3g sachets containing placebo per day - once 30-40 min before breakfast, once 30-40 min before lunch, and once 30-40 min before dinner. Participants will open the sachet, empty contents into their mouth, and let it dissolve before swallowing.
  Interventions: Drug: Fermented Papaya Preparation (FPP); Drug: Sugar Pill

INTERVENTIONS:
Drug: Fermented Papaya Preparation (FPP) — A total of 9 grams of FPP per day (divided into three 3 gram doses) will be consumed for 8 weeks. Participants will consume three 3g sachets containing FPP per day - once 30-40 min before breakfast, once 30-40 min before lunch, and once 30-40 min before dinner. Participants will open the sachet, slowly empty contents into their mouth, and let it dissolve before swallowing.
  Other Names: Papaya
Drug: Sugar Pill — A total of 9 grams of placebo (sugar) per day (divided into three 3 gram doses) will be consumed for 8 weeks. Participants will consume three 3g sachets containing placebo per day - once with breakfast, once with lunch, and once with dinner. Participants will open the sachet, empty contents into their mouth, and let it dissolve before swallowing.

SUMMARY:
The purpose of this research study is to explore the effects of fermented papaya preparation (FPP) on whole body inflammation, physical function, fatigue, and health-related quality of life. The investigators will conduct a double-blind, randomized, placebo-controlled pilot study on FPP in older adults. If FPP is found to have a beneficial impact on systematic inflammation in this study population (adults aged 70-100 years old), then this supplement may be a potential treatment option to combat aging.

DETAILED DESCRIPTION:
All of the participants in this research study will be divided randomly into one of two groups: (1) a group taking fermented papaya preparation (FPP) for 8 weeks then taking placebo for 8 weeks or (2) a group taking placebo for 8 weeks then taking FPP for 8 weeks. Placebo sachets do not contain any treatment product. Participants will be assigned randomly to be in one of these two groups.

Participants will be asked to take study product for 8 weeks each, and participation in the study will last for a total of approximately 22 weeks. Participants will be asked to attend five study visits at the University of Florida's Institute on Aging - Clinical & Translational Research Building (IOA - CTRB): Screening Visit, Visit 1, Visit 2, Visit 3, and Visit 4. Visit 1 will take place approximately 30 days after the Screening Visit. Visit 2 will take place approximately 8 weeks after the Screening Visit. Visit 3 will take place approximately 16 weeks after the Screening Visit. Visit 4 will take place approximately 20 weeks after the Screening Visit. Participants will be asked to fast (i.e., no food or liquids except water) for 8 hours prior to all clinic visits. Each visit will take approximately 1.5 to 2 hours.

Participants will also be called weekly during the study to ask how they are feel and to find out and if they remembered to take all of their study product. Finally, investigators will call approximately two weeks after participants stop taking the study product to ask how they are feeling.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 25 and < 40 kg/m2;
* Willing and able to participate in all aspects of the study;
* Self-reported sedentary to moderately active lifestyle (<120 min aerobic activity/week);
* Self-reported ability to walk ¼ mile without the use of an assistive device (i.e., cane, walker, crutch);
* Mild to Moderate physical impairment (SPPB score 4-10);
* Not confined to a wheelchair;
* Mini Mental Status Exam score > 24;
* Able to swallow study product as directed.

Exclusion Criteria:

* Failure to give consent;
* Active treatment for cancer (< 3 years);
* Stroke (< 6 mo);
* Serious heart condition, peripheral vascular disease, coronary artery disease (myocardial infarction<6 mo), Class III, IV Congestive Heart Failure;
* Severe anemia (Hgb < 8.0 g/dL);
* Liver or renal disease;
* Diabetes;
* Severe osteoarthritis;
* Fracture in upper or lower extremity within the last 6 months;
* Upper or lower extremity amputation;
* Anticoagulant therapy (aspirin use is permitted);
* Parkinson's disease;
* Severe psychiatric disease or psychological disorder (e.g., severe depression, bi-polar disorder, schizophrenia) or current use of antipsychotics;
* Current use of anabolic medications (e.g., growth hormone or testosterone) or anticholinesterase inhibitor (i.e., Aricept);
* High amounts of physical activity (i.e., running, bicycling, etc.) > 120 min/week;
* Excessive alcohol use (>2 drinks per day);
* Use of tobacco products;
* Resting heart rate > 120 bpm;
* Blood pressure with Systolic > 160mmHg and Diastolic >90mmHg;
* History of significant head injury leading to cognitive impairments;
* Visual or hearing impairments that would interfere with testing;
* Current consumption of any dietary supplements containing resveratrol, quercetin, or P. cuspidatum, grape seed extract, or ginko biloba;
* Allergies to papaya or foods with similar compounds (i.e., banana, avocado, kiwi, chestnuts, hazel nuts)
* Allergy to latex;
* Participating in another clinical trial or has received an investigational product within 30 days prior to screening/enrollment;
* Center for Epidemiological Studies - Depression Scale (CES-D) Score > 20.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) will be tested at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  Blood test performed.
Tumor necrosis factor-α (TNF-α) will be tested at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  Blood test will be performed.
C - reactive protein (CRP) will be tested at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  Blood test will be performed.
Myeloperoxidase (MPO) will be tested at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  Blood test will be performed.

SECONDARY OUTCOMES:
Short Physical Performance Battery | Change from 8 weeks and 20 weeks
  Physical function test to assess functional performance on different tasks including timed short distance walk, repeated chair stands, and a balance test.
6 Minute Walk Test performed at weeks 8 and 20. | Change from 8 weeks and 20 weeks
  The 6 Minute Walk tests functional walking endurance. Participants will be asked to walk at a comfortable pace for 6 minutes. Total distance completed, blood pressure, and pulse rate will be measured.
Health-related quality of life performed at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  RAND SF-36 Short Form Health Survey (SF-36) measures eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, vitality (energy/fatigue), emotional well being, bodily pain, social functioning, and general health perceptions.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) performed at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  FACIT-Fatigue is a measure of physical and functional consequences of fatigue, with lower scores indicating more fatigue.
Brief Fatigue Symptom Inventory (FSI) | Change from 8 weeks and 20 weeks
  FSI is a measure of physical and functional consequences of fatigue.
Superoxide dismutases (SOD) tested at weeks 8 and 20. | Change from 8 weeks and 20 weeks
  Blood test will be performed.
Glutathione Peroxidase tested at weeks 8 and 20. | Change from 8 weeks and 20 weeks
  Blood test will be performed.
Total Antioxidant Capacity will be tested at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  Blood test will be performed.
Muscle tissue oxygenation tested at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  Participants will be asked to perform a leg extension endurance exercise with electrodes placed on their forehead and thigh.
Brain tissue oxygenation tested at weeks 8 and 20 | Change from 8 weeks and 20 weeks
  Participants will complete a series of memory and thinking tasks while wearing electrodes on their head. The N-Back Test that measures working memory will be conducted for 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Anton, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States